CLINICAL TRIAL: NCT04709770
Title: Comparison of Low-volume Versus High-volume Polyethylene Glycol Based Bowel Preparation for Colonoscopy in People Receiving Hemodialysis: a Randomized Non-inferiority Trial
Brief Title: Low-volume vs High-volume Polyethylene Glycol Based Bowel Preparation for Colonoscopy in People Receiving Hemodialysis
Acronym: PrepDial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alfredo Di Leo (Other)
Collaborators: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor-Investigator, Alfredo Di Leo, Full professor, University of Bari
Organization: University of Bari (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Policlinic Hospital 7
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Chronic Kidney Diseases; Colon Polyp; Dialysis; Complications; Colon Cancer
Keywords: Colonoscopy; Bowel cleansing; Adenoma detection; Polyethylene glycol; Hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Colonic Polyps; Colonic Neoplasms | interventions — Citric Acid; Simethicone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-volume preparation (Experimental): Low-volume preparation of 2-liters polyethylene glycol with citrate and simethicone. This formulation includes 4 large (A) and 4 small (B) sachets; the components of 2 sachets A and 2 sachets B are mixed in 1 liter of water.
  Each sachet A contains:
  * polyethylene glycol (4000) 52.50 g;
  * simethicone 0.08 g;
  * sodium sulphate anhydrous 3.75 g.
  Each sachet B contains:
  * sodium citrate 1.863 g;
  * anhydrous citric acid 0.813 g;
  * sodium chloride 0.73 g;
  * potassium chloride: 0.37 g;
  * acesulfame potassium 0.13 g. Participants will drink the first liter of preparation at 19.00 p.m. on the day before the colonoscopy, at a rate of 250 ml every 15 minutes, followed by 500 ml of clear liquids. The second liter of preparation will be administered at 7.00 a.m. on the day of the colonoscopy, at a rate of 250 ml every 15 minutes, followed by 500 ml of clear liquids.
  Interventions: Drug: 2-liters polyethylene glycol with citrate and simethicone; Dietary Supplement: Low-residue diet
- High-volume preparation (Active Comparator): High-volume preparation with 4-liters polyethyleneglycol with simethicone. This formulation includes 4 sachets, each dissolved in 1 liter of water.
  Each sachet contains:
  * polyethylene glycol (4000) 58.30 g;
  * simethicone 0.08 g;
  * sodium sulphate anhydrous 5.68 g;
  * sodium bicarbonate 1.68 g;
  * sodium chloride 1.46 g;
  * potassium chloride 0.74 g. Participants will drink the first 2 liters of preparation at 19.00 p.m. on the day before colonoscopy, at a rate of 250 ml every 15 minutes. The remaining 2 liters of preparation will be administered at 6.00 a.m. on the day of the endoscopic procedure, at a rate of 250 ml every 15 minutes.
  Interventions: Drug: 4-liters polyethylene glycol with simethicone; Dietary Supplement: Low-residue diet

INTERVENTIONS:
Drug: 2-liters polyethylene glycol with citrate and simethicone — Low-volume polyethylene glycol-based bowel cleansing agent for colonoscopy.
  Other Names: Clensia
  Arms: Low-volume preparation
Drug: 4-liters polyethylene glycol with simethicone — High-volume polyethylene glycol-based bowel cleansing agent for colonoscopy.
  Other Names: Selg Esse
  Arms: High-volume preparation
Dietary Supplement: Low-residue diet — Diet before colonoscopy.

SUMMARY:
Current American Society for Gastrointestinal Endoscopy (ASGE) and European Society of Gastrointestinal Endoscopy (ESGE) guidelines recommend a split regimen of high-volume (4-liter polyethylene glycol-based preparation) or low-volume (2-liter polyethylene glycol-based solutions or sodium picosulphate plus magnesium citrate) formulations for routine bowel preparation.

Some concerns have been raised about the use of oral bowel-cleansing agents in people receiving hemodialysis due to the possibility of secondary intravascular depletion. There is a risk for thrombosis of dialysis access in case of hypotension. The association of hemodialysis treatment and the use of bowel preparations may induce severe hypovolaemia. Finally, the 4-liter intake with high-volume preparations may cause fluid overload in anuric patients.

The aim of our study will be to assess in a randomized trial the non-inferiority of a low-volume versus a high-volume polyethylene glycol-based bowel preparation for adequate bowel cleansing in people receiving hemodialysis (primary end-point). We will also compare the low-volume versus the high-volume preparation for other endoscopic and nephrologic relevant clinical outcomes (secondary end-points).

DETAILED DESCRIPTION:
Study design:

This will be a multicentre, outcome assessor-blinded, parallel-arm, centrally randomized, non-inferiority trial. Randomization will be performed centrally by the coordinating center.

Consecutive inpatients and outpatients on hemodialysis with an indication to undergo colonoscopy (positive fecal occult blood test or fecal immunochemical test, signs or symptoms of colorectal disease, colorectal cancer screening, colorectal cancer surveillance, inflammatory bowel diseases, or inclusion in kidney transplantation waiting list) will be screened for inclusion in the trial.

At enrolment visit, eligible subjects will be allocated to either the low-volume or high-volume bowel preparation group (ratio 1:1). Participants in the low-volume group will receive the formulation of 2-liters polyethylene glycol with citrate and simethicone (Clensia, Alfasigma S.p.A., Milan, Italy), while those in the high-volume arm will receive 4-liters polyethylene glycol with simethicone (Selg Esse, Alfasigma S.p.A., Milan, Italy). Participants in both groups will be prescribed a low residue diet for 3 days before colonoscopy and will be instructed to take the bowel cleansing agents as split dose, taking the first half of solution the evening before the endoscopic examination and the second in the morning of the day of the procedure. To improve compliance, participants will also receive a booklet in plain language to explain the details of low residue diet and modality of bowel preparation intake.

All endoscopic examinations will be scheduled on days free from dialysis sessions between 2 and 5 hours after the end of the administration of the last dose of preparation. On the day of the colonoscopy, all participants will fill in a questionnaire to measure participants' compliance, tolerability, and willingness to repeat the preparation they have been allocated to. Participants will be aware of the bowel preparation they received. On the opposite, endoscopists and nephrologists measuring primary and secondary outcomes (i.e. outcome assessors) will be blinded to the arm each subject has been allocated to and instructed to avoid any discussion with participants that could reveal the type of bowel cleansing agent.

Recruitment will last 12 months and follow-up will be completed 1 month after the last participant undergoes colonoscopy.

Before randomization and during the one-month follow-up, participants will receive (in a non-randomized fashion) all relevant co-interventions (e.g. iron, lipid-lowering agents, bone disease agents, antihypertensive agents, etc.), which are peculiar of standard hemodialysis treatment, as per their usual attending physician's practice to achieve and maintain standard hemodialysis clinical performance measures.

At the time of enrolment and colonoscopy scheduled simple trial follow-up visits will be performed. All clinical events following the endoscopic procedure will be measured during the one-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* prevalent end stage kidney disease on hemodialysis people (on hemodialysis for ≥6 months; either hemodialysis or hemofiltration or hemodiafiltration, received for at least 3 times/week for a minimum duration of 4 hours per treatment session for a minimum of 12 hours/week, according to standard practice for quality hemodialysis in Italy);
* inpatients and outpatients with an indication to colonoscopy (e.g. positive fecal occult blood test or fecal immunochemical test, signs or symptoms of colorectal disease, colorectal cancer screening, colorectal cancer surveillance, inflammatory bowel diseases, or inclusion in kidney transplantation waiting list);
* signature of written informed consent.

Exclusion Criteria:

* end stage kidney disease not on hemodialysis (eg. peritoneal dialysis or kidney transplantation);
* previous kidney transplantation;
* need for colonoscopy in emergency;
* previous colorectal surgery;
* contraindications to colonoscopy in the opinion of the managing physician;
* pregnancy or breastfeeding assessed by dedicated pregnancy tests;
* known or suspected hypersensitivity to any components of preparations.
* gastrointestinal perforation;
* toxic megacolon;
* inflammatory bowel disease (such as rectal ulcerative colitis, Crohn's disease) in severe acute phase;
* occlusive, sub-occlusive or stenotic forms of the intestine, gastric stasis, dynamic ileus, paralytic ileus;
* severe state of dehydration;
* phenylketonuria (due to the presence of aspartame);
* glucose-6-phosphate dehydrogenase deficiency;
* severe heart failure: New York Heart Association (NYHA) class III-IV;
* significant alterations of electrolytes, according to the physician's judgment;
* participation in a clinical study in which an experimental drug was administered within 30 days or 5 half-lives before the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Adequate bowel preparation | During colonoscopy
  Proportion of participants with Boston Bowel Preparation Scale ≥6 with each segmental score ≥2

SECONDARY OUTCOMES:
Adenoma detection rate | During colonoscopy
  Proportion of patients with at least one adenoma
Cecal intubation rate | During colonoscopy
  Proportion of endoscopic examinations reaching the cecum
Participants' compliance | During colonoscopy
  Proportion of participants with intake of at least 75 percent of the bowel preparation
Participants' tolerability | During colonoscopy
  Proportion of participants presenting nausea, bloating, vomiting, abdominal pain, and/or anal irritation
Willingness to repeat the preparation | During colonoscopy
  Proportion of participants willing to use the same bowel preparation for future examinations
Adverse events | During colonoscopy and the first hemodialysis session following colonoscopy
  Proportion of participants with any adverse event occurred during the intake of bowel preparation
All-cause hospitalization | Within a 30-day period
  Proportion of participants hospitalized after bowel preparation intake for any cause
All-cause mortality | Within a 30-day period
  Proportion of participants who died after bowel preparation intake for any cause
Emergency hemodialysis sessions | Within a 30-day period
  Proportion of participants needing additional hemodialysis sessions
Cardiovascular events | Within a 30-day period
  Proportion of participants with cardiovascular events (i.e. nonfatal myocardial infarction, acute coronary syndrome, and/or heart failure)
Interdialytic body weight gain | During the hemodialysis session preceding and the one following the intake of bowel preparation
  Mean increase in body weight from the hemodialysis session preceding the intake of bowel preparation to the one following the colonoscopy
Variations in serum-electrolyte levels | During the hemodialysis session preceding and the one following the intake of bowel preparation
  Mean variation in serum-electrolyte levels between the hemodialysis session preceding and following the intake of bowel preparation
Systolic blood pressure | During the hemodialysis session preceding and the one following the intake of bowel preparation
  Mean variation in systolic blood pressure between the hemodialysis session preceding and following the intake of bowel preparation
Diastolic blood pressure | During the hemodialysis session preceding and the one following the intake of bowel preparation
  Mean variation in diastolic blood pressure between the hemodialysis session preceding and following the intake of bowel preparation
Blood flow on dialysis | During the hemodialysis session preceding and the one following the intake of bowel preparation
  Mean variation in blood flow on dialysis between the hemodialysis session preceding and following the intake of bowel preparation

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Di Leo, MD PhD, Principal Investigator — University of Bari

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luyckx VA, Tonelli M, Stanifer JW. The global burden of kidney disease and the sustainable development goals. Bull World Health Organ. 2018 Jun 1;96(6):414-422D. doi: 10.2471/BLT.17.206441. Epub 2018 Apr 20. PMID 29904224
- [Background] de Jager DJ, Grootendorst DC, Jager KJ, van Dijk PC, Tomas LM, Ansell D, Collart F, Finne P, Heaf JG, De Meester J, Wetzels JF, Rosendaal FR, Dekker FW. Cardiovascular and noncardiovascular mortality among patients starting dialysis. JAMA. 2009 Oct 28;302(16):1782-9. doi: 10.1001/jama.2009.1488. PMID 19861670
- [Background] Komaki Y, Komaki F, Micic D, Ido A, Sakuraba A. Risk of Colorectal Cancer in Chronic Kidney Disease: A Systematic Review and Meta-Analysis. J Clin Gastroenterol. 2018 Oct;52(9):796-804. doi: 10.1097/MCG.0000000000000880. PMID 28723862
- [Background] Williams AW, Dwyer AC, Eddy AA, Fink JC, Jaber BL, Linas SL, Michael B, O'Hare AM, Schaefer HM, Shaffer RN, Trachtman H, Weiner DE, Falk AR; American Society of Nephrology Quality, and Patient Safety Task Force. Critical and honest conversations: the evidence behind the "Choosing Wisely" campaign recommendations by the American Society of Nephrology. Clin J Am Soc Nephrol. 2012 Oct;7(10):1664-72. doi: 10.2215/CJN.04970512. Epub 2012 Sep 13. PMID 22977214
- [Background] Abramowicz D, Cochat P, Claas FH, Heemann U, Pascual J, Dudley C, Harden P, Hourmant M, Maggiore U, Salvadori M, Spasovski G, Squifflet JP, Steiger J, Torres A, Viklicky O, Zeier M, Vanholder R, Van Biesen W, Nagler E. European Renal Best Practice Guideline on kidney donor and recipient evaluation and perioperative care. Nephrol Dial Transplant. 2015 Nov;30(11):1790-7. doi: 10.1093/ndt/gfu216. Epub 2014 Jul 9. PMID 25007790
- [Background] Harewood GC, Sharma VK, de Garmo P. Impact of colonoscopy preparation quality on detection of suspected colonic neoplasia. Gastrointest Endosc. 2003 Jul;58(1):76-9. doi: 10.1067/mge.2003.294. PMID 12838225
- [Background] Froehlich F, Wietlisbach V, Gonvers JJ, Burnand B, Vader JP. Impact of colonic cleansing on quality and diagnostic yield of colonoscopy: the European Panel of Appropriateness of Gastrointestinal Endoscopy European multicenter study. Gastrointest Endosc. 2005 Mar;61(3):378-84. doi: 10.1016/s0016-5107(04)02776-2. PMID 15758907
- [Background] Rex DK, Imperiale TF, Latinovich DR, Bratcher LL. Impact of bowel preparation on efficiency and cost of colonoscopy. Am J Gastroenterol. 2002 Jul;97(7):1696-700. doi: 10.1111/j.1572-0241.2002.05827.x. PMID 12135020
- [Background] ASGE Standards of Practice Committee; Saltzman JR, Cash BD, Pasha SF, Early DS, Muthusamy VR, Khashab MA, Chathadi KV, Fanelli RD, Chandrasekhara V, Lightdale JR, Fonkalsrud L, Shergill AK, Hwang JH, Decker GA, Jue TL, Sharaf R, Fisher DA, Evans JA, Foley K, Shaukat A, Eloubeidi MA, Faulx AL, Wang A, Acosta RD. Bowel preparation before colonoscopy. Gastrointest Endosc. 2015 Apr;81(4):781-94. doi: 10.1016/j.gie.2014.09.048. Epub 2015 Jan 14. No abstract available. PMID 25595062
- [Background] Hassan C, Bretthauer M, Kaminski MF, Polkowski M, Rembacken B, Saunders B, Benamouzig R, Holme O, Green S, Kuiper T, Marmo R, Omar M, Petruzziello L, Spada C, Zullo A, Dumonceau JM; European Society of Gastrointestinal Endoscopy. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) guideline. Endoscopy. 2013;45(2):142-50. doi: 10.1055/s-0032-1326186. Epub 2013 Jan 18. PMID 23335011
- [Background] Johnson DA, Barkun AN, Cohen LB, Dominitz JA, Kaltenbach T, Martel M, Robertson DJ, Boland CR, Giardello FM, Lieberman DA, Levin TR, Rex DK; US Multi-Society Task Force on Colorectal Cancer. Optimizing adequacy of bowel cleansing for colonoscopy: recommendations from the US multi-society task force on colorectal cancer. Gastroenterology. 2014 Oct;147(4):903-24. doi: 10.1053/j.gastro.2014.07.002. No abstract available. PMID 25239068
- [Background] Connor A, Tolan D, Hughes S, Carr N, Tomson C. Consensus guidelines for the safe prescription and administration of oral bowel-cleansing agents. Gut. 2012 Nov;61(11):1525-32. doi: 10.1136/gutjnl-2011-300861. Epub 2012 Jul 26. PMID 22842619
- [Background] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102
- [Background] Mahmood S, Farooqui SM, Madhoun MF. Predictors of inadequate bowel preparation for colonoscopy: a systematic review and meta-analysis. Eur J Gastroenterol Hepatol. 2018 Aug;30(8):819-826. doi: 10.1097/MEG.0000000000001175. PMID 29847488
- [Background] Hassan C, Fuccio L, Bruno M, Pagano N, Spada C, Carrara S, Giordanino C, Rondonotti E, Curcio G, Dulbecco P, Fabbri C, Della Casa D, Maiero S, Simone A, Iacopini F, Feliciangeli G, Manes G, Rinaldi A, Zullo A, Rogai F, Repici A. A predictive model identifies patients most likely to have inadequate bowel preparation for colonoscopy. Clin Gastroenterol Hepatol. 2012 May;10(5):501-6. doi: 10.1016/j.cgh.2011.12.037. Epub 2012 Jan 10. PMID 22239959
- [Background] The Paris endoscopic classification of superficial neoplastic lesions: esophagus, stomach, and colon: November 30 to December 1, 2002. Gastrointest Endosc. 2003 Dec;58(6 Suppl):S3-43. doi: 10.1016/s0016-5107(03)02159-x. No abstract available. PMID 14652541
- [Background] Kang X, Zhao L, Zhu Z, Leung F, Wang L, Wang X, Luo H, Zhang L, Dong T, Li P, Chen Z, Ren G, Jia H, Guo X, Pan Y, Guo X, Fan D. Same-Day Single Dose of 2 Liter Polyethylene Glycol is Not Inferior to The Standard Bowel Preparation Regimen in Low-Risk Patients: A Randomized, Controlled Trial. Am J Gastroenterol. 2018 Apr;113(4):601-610. doi: 10.1038/ajg.2018.25. Epub 2018 Mar 13. PMID 29533397
- [Background] Kump P, Hassan C, Spada C, Brownstone E, Datz C, Haefner M, Renner F, Schoefl R, Schreiber F. Efficacy and safety of a new low-volume PEG with citrate and simethicone bowel preparation for colonoscopy (Clensia): a multicenter randomized observer-blind clinical trial vs. a low-volume PEG with ascorbic acid (PEG-ASC). Endosc Int Open. 2018 Aug;6(8):E907-E913. doi: 10.1055/a-0624-2266. Epub 2018 Aug 1. PMID 30083580
- [Background] Spada C, Cesaro P, Bazzoli F, Saracco GM, Cipolletta L, Buri L, Crosta C, Petruzziello L, Ceroni L, Fuccio L, Giordanino C, Elia C, Rotondano G, Bianco MA, Simeth C, Consalvo D, De Roberto G, Fiori G, Campanale M, Costamagna G. Evaluation of Clensia(R), a new low-volume PEG bowel preparation in colonoscopy: Multicentre randomized controlled trial versus 4L PEG. Dig Liver Dis. 2017 Jun;49(6):651-656. doi: 10.1016/j.dld.2017.01.167. Epub 2017 Feb 3. PMID 28233684
- [Result] Lee JM, Keum B, Yoo IK, Kim SH, Choi HS, Kim ES, Seo YS, Jeen YT, Chun HJ, Lee HS, Um SH, Kim CD, Kim MG, Jo SK. Polyethylene glycol plus ascorbic acid for bowel preparation in chronic kidney disease. Medicine (Baltimore). 2016 Sep;95(36):e4755. doi: 10.1097/MD.0000000000004755. PMID 27603372
- [Result] Yoshida N, Naito Y, Murakami T, Hirose R, Ogiso K, Inada Y, Dohi O, Okayama T, Kamada K, Uchiyama K, Ishikawa T, Handa O, Konishi H, Siah KT, Yagi N, Itoh Y. Safety and Efficacy of a Same-Day Low-Volume 1 L PEG Bowel Preparation in Colonoscopy for the Elderly People and People with Renal Dysfunction. Dig Dis Sci. 2016 Nov;61(11):3229-3235. doi: 10.1007/s10620-016-4262-7. Epub 2016 Aug 3. PMID 27487795